CLINICAL TRIAL: NCT06575192
Title: A Prospective, Multicenter, Open-Label, Non-Randomized, Controlled Pivotal Study to Evaluate the Safety and Effectiveness of ARTIA Reconstructive Tissue Matrix in Implant-Based Two Stage Prepectoral Breast Reconstruction Post-Mastectomy
Brief Title: Evaluation of the Safety and Effectiveness of ARTIA Reconstructive Tissue Matrix Breast Reconstruction (ADORA) in Adult Participants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-708
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Reconstruction
Keywords: Breast Reconstruction; ADORA; ARTIA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acellular Dermal Matrix (Experimental): Breast reconstruction with ARTIA Tissue Matrix.
  Interventions: Device: ARTIA Reconstructive Tissue Matrix
- Non-Acellular Dermal Matrix (ADM) Control Group (Other): Breast reconstruction without ADM.
  Interventions: Other: No Intervention

INTERVENTIONS:
Device: ARTIA Reconstructive Tissue Matrix — Surgical Implant
  Arms: Acellular Dermal Matrix
Other: No Intervention — No ADM
  Arms: Non-Acellular Dermal Matrix (ADM) Control Group

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of ARTIA in adult participants undergoing immediate, two-stage, implant-based breast reconstruction post-mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will undergo unilateral or bilateral mastectomy upon enrollment.
* Participants who are willing and able to undergo immediate pre-pectoral two-stage breast reconstruction with ARTIA or without ADM.

Exclusion Criteria:

* Has an existing carcinoma of the breast without planned mastectomy or residual gross local tumor of the breast after mastectomy.
* Has any disease which is clinically known to impact wound healing ability, such as uncontrolled diabetes or history of compromised wound healing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 783 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of at Least One Major Complication related to Breast Reconstruction After Stage 1 | Month 18
  Number of participants with at least one major complication related to breast reconstruction.
Change from Baseline in BREAST-Q Satisfaction with Breasts Score from Pre-Mastectomy After Stage 2 | Up to Month 18
  Participants evaluated satisfaction with their breasts using the BREAST-Q. Summary scores were computed by summing the score of each response and transferring them to a 0 (worst) to 100 (best) scale.
Number of Participants with Adverse Events (AEs) | Up to Approximately 36 Months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a medical device which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Occurrence of Capsular Contracture per Breast | Month 36
  Number of participants with an occurrence of capsular contracture per breast.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (20):
- United States (20):
  - Cedars-Sinai Medical Center /ID# 268326, Los Angeles, California
  - UC Irvine Medical Center /ID# 267428, Orange, California
  - Stanford University Medical Center CTRU - 800 Welch Road /ID# 264196, Palo Alto, California
  - South Bay Plastic Surgeons /ID# 264192, Torrance, California
  - University Of Colorado - Anschutz Medical Campus /ID# 268627, Aurora, Colorado
  - University of Florida College of Medicine /ID# 267485, Gainesville, Florida
  - Endeavor Health /ID# 266302, Northbrook, Illinois
  - Johns Hopkins Hospital /ID# 265917, Baltimore, Maryland
  - Washington University School of Medicine - St. Louis /ID# 264029, St Louis, Missouri
  - University of Nevada - Main Campus /ID# 264017, Las Vegas, Nevada
  - Rutgers New Jersey Medical School - Newark /ID# 264187, Newark, New Jersey
  - Northwell Health Clinical Trials Office /ID# 268076, Lake Success, New York
  - NYU Langone Medical Center /ID# 265621, New York, New York
  - Atrium Health Wake Forest Baptist Medical Center /ID# 264382, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center /ID# 266253, Columbus, Ohio
  - Erlanger Health System /ID# 266608, Chattanooga, Tennessee
  - East Tennessee State University /ID# 264321, Johnson City, Tennessee
  - The University of Texas MD Anderson Cancer Center /ID# 264020, Houston, Texas
  - University of Virginia /ID# 265098, Charlottesville, Virginia
  - AG Aesthetic Center /ID# 264233, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-708